CLINICAL TRIAL: NCT01334320
Title: Survival Benefit of Elective Neck Dissection for Patients With T1,2N0M0 Oral Squamous Cell Carcinoma-A Prospective Multicenter Randomized Controlled Study
Brief Title: Survival Benefit of Elective Neck Dissection in T1,2N0M0 Oral Squamous Cell Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Gui-Qing Liao, Guanghua School of Stomatology, Hospital of Stomatology, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010018
Record Dates: First submitted 2011-04-06; First posted 2011-04-13 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Oral Squamous Cell Carcinoma
Keywords: oral squamous cell carcinoma; elective neck dissection; "watchful waiting"; survival benefit; recurrence rate
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- elective neck dissection (Experimental): patient underwent elective neck dissection as initial treatment, along with the excision of the primary tumor
  Interventions: Procedure: elective neck dissection
- wait and see (No Intervention): patient underwent primary tumor excision transorally as initial treatment, and without a cervical intervention

INTERVENTIONS:
Procedure: elective neck dissection — patient underwent elective neck dissection as initial treatment, along with the excision of the primary tumor
  Other Names: superior omohyoid neck dissection, SOHND
  Arms: elective neck dissection

SUMMARY:
Controversy over surgical treatment of clinically negative neck in early stage oral squamous cell carcinoma revolves around the uncertainty of its impact on patient prognosis. The efficacy of elective neck dissection on prognosis in T1, 2 N0M0 patients continues to be the subject of clinical debate. Currently the clinically negative patients are treated by one of the two main policies: one is elective neck dissection; the other is "watchful waiting". The objective of this multi-institutional prospective randomized controlled study is to evaluate the survival benefit of elective neck dissection on the prognosis of T1, 2 N0M0 patients with carcinoma of oral cavity. The enrolled patients with T1, 2 N0M0 oral cancer will be randomized into two groups: elective neck dissection versus watch and wait. The survival rate and the recurrence rate between two groups will be compared. The result of the study will give surgeons evidence-based instructions for the management of clinically negative neck in patients with cancer of oral cavity.

DETAILED DESCRIPTION:
There are controversies on the benefits of elective neck dissection (END) for clinically negative neck in early stage oral squamous cell carcinoma. The aim of this study is to determine the need for a randomized controlled trial in order to evaluate the survival benefit of elective neck dissection on the prognosis of T1, 2 N0M0 patients with carcinoma of oral cavity. We initiate this multi-institutional study, expecting 448 primary oral cancer patients to be enrolled. And we are going to randomly divide these patients into two groups: END and "watch and wait". The END group will undergo one stage surgery of END and primary tumor excision, and the "watch and wait"group will be treated with primary tumor excision transorally as initial treatment, with rigorous postoperation consultation. All patients will be followed up with at least 5 years after initial treatment, and the survival rate and the recurrence rate between groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Age:20 to 70 years old, both male and female
2. Histologically proven T1 or T2 N0 M0 (clinical) squamous cell carcinoma of the oral tongue, buccal mucosa, gingiva, floor of mouth, and hard palate
3. The maximum diameter of the primary tumor is less than 4cm
4. Clinical nodal staging has been confirmed negative via both clinical examination and imaging (MRI or lateral and central neck ultrasound)
5. With at least 1-year's expected survival time
6. Willing to join the protocol and is able to give written informed consent

Exclusion Criteria:

1. Patient with severe cardiac insufficiency, hepatic insufficiency, renal insufficiency, of systemic infection diseases
2. The patient is pregnant or lactating
3. Patients with a history of surgical treatment, radiotherapy, chemotherapy, biotherapy and targeted therapy, et al, before participating in the study
4. Patient is currently participating in another investigational drug study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Estimated)
Dates: Start 2011-04; Primary Completion 2015-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Whether elective neck dissection (END) has equal or higher survival rate to the wait and watch policy | 5 years
  The 5-year's survival and the disease free survival of the two group of patients are being measured and compared with one and other, so the survival benefit of the two policy is evaluated.

SECONDARY OUTCOMES:
Does END have the equal or lower recurrence rate to the wait and watch policy | 5 years
  The recurrence includes recurrence of the primary tumor and the neck, and it's measured by clinical examination, MRI examination and ultrasonic inspection.
quality of life | 5 years
  The quality of life of patients after surgery is measured by UW-QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Guiqing Liao, MD, DDS, Principal Investigator — Sun Yat-sen University
Locations (4):
- China (4):
  - Hospital of Stomatology, Sun Yat-sen University, Guangzhou, Guangdong
  - Cancer Center, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong

REFERENCES:
- [Background] Yuen AP, Ho CM, Chow TL, Tang LC, Cheung WY, Ng RW, Wei WI, Kong CK, Book KS, Yuen WC, Lam AK, Yuen NW, Trendell-Smith NJ, Chan YW, Wong BY, Li GK, Ho AC, Ho WK, Wong SY, Yao TJ. Prospective randomized study of selective neck dissection versus observation for N0 neck of early tongue carcinoma. Head Neck. 2009 Jun;31(6):765-72. doi: 10.1002/hed.21033. PMID 19408291
- [Background] D'Cruz AK, Siddachari RC, Walvekar RR, Pantvaidya GH, Chaukar DA, Deshpande MS, Pai PS, Chaturvedi P. Elective neck dissection for the management of the N0 neck in early cancer of the oral tongue: need for a randomized controlled trial. Head Neck. 2009 May;31(5):618-24. doi: 10.1002/hed.20988. PMID 19132717
- [Background] Rodrigo JP, Shah JP, Silver CE, Medina JE, Takes RP, Robbins KT, Rinaldo A, Werner JA, Ferlito A. Management of the clinically negative neck in early-stage head and neck cancers after transoral resection. Head Neck. 2011 Aug;33(8):1210-9. doi: 10.1002/hed.21505. Epub 2010 Dec 6. PMID 21755564
- [Derived] Worthington HV, Bulsara VM, Glenny AM, Clarkson JE, Conway DI, Macluskey M. Interventions for the treatment of oral cavity and oropharyngeal cancers: surgical treatment. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD006205. doi: 10.1002/14651858.CD006205.pub5. PMID 37650478
- See also: citation 3 — http://www.ncbi.nlm.nih.gov/pubmed/?term=Management+of+the+clinically+negative+neck+in+early-stage+head+and+neck+cancers+after+transoral+resection
- See also: citation 2 — http://www.ncbi.nlm.nih.gov/pubmed/?term=Elective+neck+dissection+for+the+management+of+the+N0+neck+in+early+cancer+of+the+oral+tongue%3A+need+for+a+randomized+controlled+trial
- See also: citation 1 — http://www.ncbi.nlm.nih.gov/pubmed/?term=Prospective+randomized+study+of+selective+neck+dissection+versus+observation+for+N0+neck+of+early+tongue+carcinoma.